CLINICAL TRIAL: NCT03601117
Title: Accelerated Intermittent Theta Burst Stimulation for Depressive Symptoms
Acronym: aTBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Nolan R, Assistant Professor, Director, Interventional Psychiatry Clinical Research, Director, Brain Stimulation Laboratory, Department of Psychiatry and Behavioral Sciences, Stanford School of Medicine, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 41071
Record Dates: First submitted 2018-07-06; First posted 2018-07-26 (Actual); Results first posted 2021-08-10 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-04

CONDITIONS: Depression and Suicide
MeSH Terms: conditions — Depression; Suicide

STUDY DESIGN:
Intervention Model Description: A small pilot study (n=22) will be an open-label study in which all participants receive stimulation to the L-DLPFC to demonstrate feasibility of delivering this accelerated protocol on an inpatient unit.
  For participants who do not respond to L-DLPFC stimulation, we will offer an alternative site, the ACC.
  If patients are enrolled that have a psychiatric diagnosis other than MDD, scales measuring symptoms related to their other diagnosis/(es) will also be collected in addition to measuring change in depressive symptoms (see 'other pre-specified outcome measures' for a list of measures used to measure symptoms related to psychiatric diagnoses other than depression).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Dorsolateral Prefrontal Cortex (Experimental): The accelerated theta burst stimulation protocol will be applied to the left dorsolateral prefrontal cortex (L-DLPFC), for 10 sessions per day for up to 5 days.
  Interventions: Device: Dorsolateral Prefrontal Cortex Accelerated Theta Burst Stimulation
- Anterior Cingulate Cortex (Experimental): The accelerated theta burst stimulation protocol will be applied to the left anterior cingulate cortex (ACC), for 10 sessions per day for up to 5 days.
  Interventions: Device: Anterior Cingulate Cortex Accelerated Theta Burst Stimulation

INTERVENTIONS:
Device: Dorsolateral Prefrontal Cortex Accelerated Theta Burst Stimulation — Participants will receive iTBS (intermittent theta burst stimulation) to the left DLPFC.
  Stimulation intensity will be standardized at 80% of resting motor threshold (adjusted for cortical depth).
  Stimulation will be delivered using the Brainsway TMS system.
  Arms: Dorsolateral Prefrontal Cortex
Device: Anterior Cingulate Cortex Accelerated Theta Burst Stimulation — Participants will receive iTBS (intermittent theta burst stimulation) to the anterior cingulate cortex (ACC).
  Stimulation intensity will be standardized at 80% of resting motor threshold (adjusted for cortical depth).
  Stimulation will be delivered using the Brainsway TMS system.
  Arms: Anterior Cingulate Cortex

SUMMARY:
This study evaluates an accelerated schedule of theta-burst stimulation for depressive symptoms in psychiatric inpatients.

A small pilot study (n=22) will be carried out to demonstrate feasibility, using the FDA-approved stimulation site for depression treatment (L-DLPFC). Participants will be offered stimulation at the anterior cingulate cortex (ACC).

DETAILED DESCRIPTION:
This study intends to investigate whether modifying stimulation parameters enables typical 6-8 week long rTMS protocols to be compressed to only five days. The influence of this accelerated protocol on the length of patient stay in the hospital will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Able to read, understand, and provide written, dated informed consent prior to screening. Participants will be deemed likely to comply with study protocol and communicate with study personnel about adverse events and other clinically important information.
* Currently diagnosed with Major Depressive Disorder (MDD) and/or in a current major depressive episode, according to the criteria defined in the Diagnosis and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR)
* Currently an inpatient at Stanford Hospital
* Meet the threshold on the total HAMD17 score of >/=20 at screening/baseline.
* Qualifies and has access to outpatient rTMS treatment

Exclusion Criteria:

* Any structural lesion e.g. structural neurological condition, more subcortical lesions than would be expected for age, stroke effecting stimulated area or connected areas or any other clinically significant abnormality that might affect safety, study participation, or confound interpretation of study results.
* Metal implant in brain (e.g. deep brain stimulation), cardiac pacemaker, or cochlear
* History of epilepsy/ seizures (including history of withdrawal/ provoked seizures)
* Shrapnel or any ferromagnetic item in the head
* Pregnancy
* Autism Spectrum disorder
* Active substance use (<1 week) or intoxication verified by toxicology screen--of cocaine, amphetamines, benzodiazepines
* Any current or past history of any physical condition which in the investigator's opinion might put the subject at risk or interfere with study results interpretation
* Cognitive impairment (including dementia)
* Current severe insomnia (must sleep a minimum of 4 hours the night before stimulation)
* Current mania
* Current unmanageable psychosis
* IQ <70
* Showing symptoms of withdrawal from alcohol or benzodiazepines
* Parkinsonism or other movement d/o determined by PI to interfere with treatment
* More subcortical lesions than would be expected for age or a stroke effecting stimulated area or connected areas.
* Any other indication the PI feels would comprise data.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nolan Williams, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] George MS, Lisanby SH, Avery D, McDonald WM, Durkalski V, Pavlicova M, Anderson B, Nahas Z, Bulow P, Zarkowski P, Holtzheimer PE 3rd, Schwartz T, Sackeim HA. Daily left prefrontal transcranial magnetic stimulation therapy for major depressive disorder: a sham-controlled randomized trial. Arch Gen Psychiatry. 2010 May;67(5):507-16. doi: 10.1001/archgenpsychiatry.2010.46. PMID 20439832
- [Background] George MS, Wassermann EM, Williams WA, Callahan A, Ketter TA, Basser P, Hallett M, Post RM. Daily repetitive transcranial magnetic stimulation (rTMS) improves mood in depression. Neuroreport. 1995 Oct 2;6(14):1853-6. doi: 10.1097/00001756-199510020-00008. PMID 8547583
- [Background] Pascual-Leone A, Rubio B, Pallardo F, Catala MD. Rapid-rate transcranial magnetic stimulation of left dorsolateral prefrontal cortex in drug-resistant depression. Lancet. 1996 Jul 27;348(9022):233-7. doi: 10.1016/s0140-6736(96)01219-6. PMID 8684201

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were recruited from Stanford Hospital
Pre-assignment Details: 23 participants signed informed consent; 22 participants were allocated to a treatment group.
Groups:
- Anterior Cingulate Cortex (ACC): The accelerated theta burst stimulation protocol will be applied to the anterior cingulate cortex (ACC), for 10 sessions per day for up to 5 days.
Period: Overall Study
Arm/Group | Dorsolateral Prefrontal Cortex | Anterior Cingulate Cortex (ACC)
Started | 20 | 2
Completed | 17 | 1
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dorsolateral Prefrontal Cortex | Anterior Cingulate Cortex (ACC) | Total
Number analyzed (Participants) | 20 | 2 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 1 | 17
  >=65 years | 4 | 1 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.55 (17.41) | 68.5 (13.44) | 47.64 (18.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 1 | 8
  Male | 13 | 1 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Non-Hispanic or Latino | 18 | 2 | 20
  Ethnicity: Hispanic or Latino | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 20 | 2 | 22
Baseline MADRS [Mean (Standard Deviation); unit: score on a scale] — A 10-item clinician-administered scale, designed to be particularly sensitive to antidepressant treatment effects in patients with major depression. Severity gradations for the MADRS have been proposed: 9-17 = mild depression, 18-34 = moderate depression, and ≥ 35 = severe depression. Scores range from 0-60.
  score on a scale | 38.5 (6.33) | 29.5 (.71) | 37.68 (6.61)

OUTCOME MEASURES:

1. Primary Outcome: Change in Montgomery Asberg Depression Rating Scale (MADRS) Score
Description: A 10-item clinician-administered scale, designed to be particularly sensitive to antidepressant treatment effects in patients with major depression. Severity gradations for the MADRS have been proposed: 9-17 = mild depression, 18-34 = moderate depression, and ≥ 35 = severe depression. Scores range from 0-60 (higher scores are more symptomatic).
  Response is defined as a 50% reduction or greater in MADRS score compared to baseline. Remission is defined as a MADRS score of <10.
  Data are presented as a raw score point change.
Time Frame: After all stimulation sessions have been completed (approximately 48 hours after the final session)
Population: Only participants who completed the protocol were included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Dorsolateral Prefrontal Cortex (L-DLPFC): The accelerated theta burst stimulation protocol will be applied to the left dorsolateral prefrontal cortex (L-DLPFC), for 10 sessions per day for up to 5 days.
Arm/Group | Dorsolateral Prefrontal Cortex (L-DLPFC) | Anterior Cingulate Cortex (ACC)
Number analyzed (Participants) | 17 | 1
score on a scale | 26.59 (10.32) | 16 (0)
Statistical Analysis 1: Comparison: Dorsolateral Prefrontal Cortex (L-DLPFC); Test type: Other — This is to test for the antidepressant effect of LDLPFC stimulation. Test is change in score from baseline to approximately 48 hours after the final session; p < .001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change in Scale of Suicidal Ideation (SSI) Score
Description: 19-item clinician administered assessment to measure the intensity, pervasiveness, and characteristics of suicidal ideation in adults.
  Scores range from 0-38. Higher scores indicate more suicidality.
  Data are presented as a raw score point change.
Time Frame: After all stimulation sessions have been completed (approximately 48 hours after the final session)
Population: Only participants who completed the questionnaire were included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Anterior Cingulate Cortex: The accelerated theta burst stimulation protocol will be applied to the anterior cingulate cortex (ACC), for 10 sessions per day for up to 5 days.
Arm/Group | Dorsolateral Prefrontal Cortex | Anterior Cingulate Cortex
Number analyzed (Participants) | 17 | 1
score on a scale | 9.82 (9.69) | 0

3. Secondary Outcome: Change in Hamilton Rating Scale for Depression Six Item (HAMD-6) Score
Description: Clinical assessment measuring depressive symptoms. Scores range from 0-24 with scores >5 indicating clinical levels of depressive symptoms (higher scores are more symptomatic).
  Data are presented as a raw score point change.
Time Frame: After all stimulation sessions have been completed (approximately 48 hours after the final session)
Population: Only participants who completed the protocol were included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dorsolateral Prefrontal Cortex | Anterior Cingulate Cortex (ACC)
Number analyzed (Participants) | 17 | 1
score on a scale | 10 (4.03) | 1 (0)

4. Secondary Outcome: Change in Young Mania Rating Scale (YMRS)
Description: The Young Mania Rating Scale (YMRS) is one of the most frequently utilized rating scales to assess manic symptoms. The scale has 11 items and is based on the patient's subjective report of his or her clinical condition.
  There are four items that are graded on a 0 to 8 scale (irritability, speech, thought content, and disruptive/aggressive behavior), while the remaining seven items are graded on a 0 to 4 scale. These four items are given twice the weight of the others to compensate for poor cooperation from severely ill patients.
  Typical YMRS baseline scores can vary a lot. They depend on the patients' clinical features such as mania (YMRS = 12), depression (YMRS = 3), or euthymia (YMRS = 2).
  Data are presented as a raw score point change.
Time Frame: After all stimulation sessions have been completed (approximately 48 hours after the final session)
Population: Only participants who completed the protocol were included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dorsolateral Prefrontal Cortex | Anterior Cingulate Cortex (ACC)
Number analyzed (Participants) | 17 | 1
score on a scale | .06 (.43) | 0 (0)

5. Secondary Outcome: Change in Beck Depression Inventory II (BDI-II)
Description: The Beck Depression Inventory (BDI-II) is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression. BDI-II items are rated on a 4-point scale ranging from 0 to 3 based on severity of each item. The maximum total score is 63.
  Scores: 0-13= minimal depression, 14-19=mild depression, 20-28=moderate depression, 29-63=severe depression.
  Data are presented as a raw score point change.
Time Frame: After all stimulation sessions have been completed (approximately 48 hours after the final session)
Population: Only participants who completed the questionnaire were included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dorsolateral Prefrontal Cortex | Anterior Cingulate Cortex (ACC)
Number analyzed (Participants) | 16 | 1
score on a scale | 18.88 (10.76) | 6 (0)

6. Secondary Outcome: Change in Quick Inventory Depressive Scale-Self Reported (QIDS) Score
Description: Self-report measure of depressive symptoms. The questionnaire consists of 16 questions. Each question can score between 0 to 4 points.
  Severity of depression is determined as follows: 0=None, 1=Mild, 2=Moderate, 3=Severe, 4=Very Severe.
  Total scores range from 0-27. Total scores: 0-5= no depression, 6-10= mild depression, 11-15= moderate depression, 16-20= severe depression, 21-27= very severe depression.
  The total score is obtained by adding the scores for each of the nine symptom domains of the DSM-IV MDD criteria: depressed mood, loss of interest or pleasure, concentration/decision making, self-outlook, suicidal ideation, energy/fatigability, sleep, weight/appetite change, and psychomotor changes (Rush et al. 2003).
  Data are presented as a raw score point change.
Time Frame: After all stimulation sessions have been completed (approximately 48 hours after the final session)
Population: Only participants who completed the protocol were included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dorsolateral Prefrontal Cortex | Anterior Cingulate Cortex (ACC)
Number analyzed (Participants) | 17 | 1
score on a scale | 11.29 (5.81) | 6 (0)

7. Secondary Outcome: Change in Pittsburgh Insomnia Rating Scale-20 Item Version (PIRS-20) Score
Description: Self-report, 20 item scale to determine patient's insomnia level.
  Each question can be scored between 0-3. 0=not bothered at all
  slightly bothered moderately bothered severely bothered
  Total score is calculated by adding up all questions (i.e. Q1+Q2+...Q20). One missing item is allowed, pro-rate if missing one item....i.e. (sum/count)*20.
  Minimum Score = 0 (good); Maximum Score = 60 (bad).
  Data are presented as a raw score point change.
Time Frame: After all stimulation sessions have been completed (approximately 48 hours after the final session)
Population: Participants who completed this questionnaire were included in the analysis. Participants who do not have this data completed were excluded.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dorsolateral Prefrontal Cortex | Anterior Cingulate Cortex (ACC)
Number analyzed (Participants) | 13 | 1
score on a scale | 16.23 (13.92) | 24 (0)

8. Secondary Outcome: Change in Resting-state Recordings and TMS-evoked Potentials in EEG Data.
Description: For the first and last stimulation session, EEG recording will be made before (resting-state EEG) and during (TMS-evoked potentials) the stimulation.
Time Frame: After all stimulation sessions have been completed (approximately 48 hours after the final session)
Population: EEG data were not collected.
Arm/Group | Dorsolateral Prefrontal Cortex (L-DLPFC) | Anterior Cingulate Cortex (ACC)
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Biomarker Analysis in Patient Blood (Plasma) Samples
Description: Blood (plasma) samples will be collected before and one month after stimulation. Blood collection is conducted by the registered hospital phlebotomist (following same protocol of a routine blood test).
  Blood samples will be analyzed by our collaborators at the Open Medicine Institute. Specifically, samples will be used for DNA/RNA extraction and analyses will be done to determine potential gene targets. Presence of inflammatory markers (cytokines) will also be determined.
  All analyses of blood samples will be conducted in the Open Medicine Institute.
Time Frame: After all stimulation sessions have been completed (approximately 48 hours after the final session)
Population: Blood samples were not collected.
Arm/Group | Dorsolateral Prefrontal Cortex | Anterior Cingulate Cortex (ACC)
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Biomarker Analysis in Patient Stool Samples
Description: Stool samples will be collected before and one month after stimulation. Stool collection is performed by registered hospital nurses.
  Stool samples will be analyzed by our collaborators at the Open Medicine Institute. Specifically, stool samples will be analyzed for potential biomarkers in the gut microbiome.
  All analyses of stool samples will be conducted in the Open Medicine Institute.
Time Frame: After all stimulation sessions have been completed (approximately 48 hours after the final session)
Population: Stool samples were not collected.
Arm/Group | Dorsolateral Prefrontal Cortex (L-DLPFC) | Anterior Cingulate Cortex (ACC)
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Biomarker Analysis in Patient Saliva Samples
Description: Saliva samples will be collected before and one month after stimulation. Saliva collection is performed by registered study personnel.
  Saliva samples will be analyzed by our collaborators at the Open Medicine Institute. Specifically, saliva samples will be analyzed for cortisol levels.
  All analyses of stool samples will be conducted in the Open Medicine Institute.
Time Frame: After all stimulation sessions have been completed (approximately 48 hours after the final session)
Population: Salvia samples were not collected.
Arm/Group | Dorsolateral Prefrontal Cortex (L-DLPFC) | Anterior Cingulate Cortex (ACC)
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Change in th Quality of Life Enjoyment and Satisfaction Questionnaire-short Form Score
Description: 15-item self-report questionnaire where each item is scored from very poor=1 to very good=5.
  The scoring of the Q-LES-Q-SF involves summing only the first 14 items to yield a raw total score.
  The last two items are not included in the total score but are stand-alone items.
  The raw total score ranges from 14 (min) to 70 (max).
Time Frame: After all stimulation sessions have been completed (approximately 48 hours after the final session)
Population: Only participants who completed this questionnaire were included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dorsolateral Prefrontal Cortex | Anterior Cingulate Cortex (ACC)
Number analyzed (Participants) | 11 | 1
score on a scale | 12.36 (13.41) | 5 (0)

13. Secondary Outcome: Change in Performance on the NIH Toolbox
Description: Neurocognitive assessments delivered through an iPad app
Time Frame: After all stimulation sessions have been completed (approximately 48 hours after the final session)
Population: NIH toolbox data was not collected.
Arm/Group | Dorsolateral Prefrontal Cortex (L-DLPFC) | Anterior Cingulate Cortex (ACC)
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Change in Immediate Mood Scaler (Ims-12) Depression Subscale Score
Description: Immediate Mood Scaler (IMS) is a newly developed, iPad-deliverable 12-item self-report tool designed to capture current mood states with overall score, and depression and anxiety subscales. Individual item scores range from 1-7, with a total overall score range from 12-84.
  Data are presented as a raw score point change in depression subscale score. The depression subscale scores range from 7-49 (higher score indicating worse depression).
Time Frame: After all stimulation sessions have been completed (approximately 48 hours after the final session)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dorsolateral Prefrontal Cortex | Anterior Cingulate Cortex (ACC)
Number analyzed (Participants) | 15 | 1
score on a scale | 11 (12.67) | -6 (0)

15. Secondary Outcome: Change in Heart Rate Variability
Description: Measure presence of any change in heart rate variability.
  Data is reported as a ratio of low frequency (LF) and high frequency (HF) (LF/HF FFT).
  FFT: fast Fourier transform.
Time Frame: After all stimulation sessions have been completed (approximately 48 hours after the final session)
Population: The device used to collect pilot HRV data was only acquired after the ACC participants had been run. Only participants with collected HRV data were included in the analysis.
Measure: Mean (Standard Deviation); unit: LF/HF FFT ratio
Arm/Group | Dorsolateral Prefrontal Cortex | Anterior Cingulate Cortex (ACC)
Number analyzed (Participants) | 3 | 0
LF/HF FFT ratio | -1.88 (3.01) |

16. Other Pre Specified Outcome: Change in Alcohol Craving Questionnaire Score (Adapted for All Drug Use)
Description: If participants have a co-morbid diagnosis of drug abuse this self-report questionnaire will be used to monitor craving of their particular drug of abuse.
Time Frame: After all stimulation sessions have been completed (approximately 48 hours after the final session)
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Change in Borderline Evaluation Of Severity Over Time (BEST) Score
Description: If participants have a co-morbid diagnosis of borderline personality disorder this self-report questionnaire will be used to monitor symptoms.
Time Frame: After all stimulation sessions have been completed (approximately 48 hours after the final session)
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Change in Obsessive Compulsive Drinking Scale Score (Adapted for Use of Any Drug)
Description: If participants have a co-morbid diagnosis of drug abuse this self-report questionnaire will be used.
Time Frame: After all stimulation sessions have been completed (approximately 48 hours after the final session)
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Change in Average Weekly Substance Use
Description: If participants have a co-morbid diagnosis of drug abuse their reported average weekly substance use will be recorded.
Time Frame: After all stimulation sessions have been completed (approximately 48 hours after the final session)
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Change in Eating Disorder Examination Questionnaire (EDE-Q) Score
Description: If participants have a co-morbid diagnosis of an eating disorder, this self-report questionnaire will be used to monitor symptoms.
Time Frame: After all stimulation sessions have been completed (approximately 48 hours after the final session)
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Change in Generalized Anxiety Disorder 7-item (GAD-7) Score
Description: If participants have a co-morbid diagnosis of Anxiety, this self-report scale will be used to monitor anxiety symptoms.
Time Frame: After all stimulation sessions have been completed (approximately 48 hours after the final session)
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Change in Yale Brown Cornell Eating Disorder Scale (YBC-EDS) Score
Description: If participants have a co-morbid diagnosis of an eating disorder, this clinician-rated assessment will be used to monitor symptoms.
Time Frame: After all stimulation sessions have been completed (approximately 48 hours after the final session)
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Change in Massachusetts General Hospital (MGH) Hairpulling Scale Score (Edited so Can be Used With Any Impulse Disorder)
Description: If participants have a co-morbid diagnosis of an impulse disorder, this self-report questionnaire will be used to monitor symptoms.
Time Frame: After all stimulation sessions have been completed (approximately 48 hours after the final session)
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Change in Obsessive Compulsive Inventory (OCI) Score
Description: If participants have a co-morbid diagnosis of OCD, this self-report questionnaire will be used to monitor symptoms.
Time Frame: After all stimulation sessions have been completed (approximately 48 hours after the final session)
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Change in Yalebrown Obsessive Compulsive Scale (YBOCS) Score
Description: If participants have a co-morbid diagnosis of OCD, this clinician-rated scale will be used to monitor symptoms.
Time Frame: After all stimulation sessions have been completed (approximately 48 hours after the final session)
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Change in Numeric Rating Scale For Pain Score
Description: If participants have a co-morbid diagnosis of a pain disorder, this rating scale will be used to monitor symptoms.
Time Frame: After all stimulation sessions have been completed (approximately 48 hours after the final session)
Reporting Status: Not Posted

27. Other Pre Specified Outcome: Change in Panic Disorder Severity Scale (PDSS) Score
Description: If participants have a co-morbid diagnosis of a panic disorder, this rating scale will be used to monitor symptoms.
Time Frame: Pre-treatment, after each day of stimulation and immediate post-treatmentAfter all stimulation sessions have been completed (approximately 48 hours after the final session)
Reporting Status: Not Posted

28. Other Pre Specified Outcome: PTSD Checklist Civilian Version (PCL-C)
Description: If participants have a co-morbid diagnosis of PTSD, this self-report questionnaire will be used to monitor symptoms.
Time Frame: After all stimulation sessions have been completed (approximately 48 hours after the final session)
Reporting Status: Not Posted

29. Other Pre Specified Outcome: Change in Calgary Depression Scale For Schizophrenia (CDSS) Score
Description: If participants have a co-morbid diagnosis of Schizophrenia, this assessment will be used to monitor symptoms.
Time Frame: After all stimulation sessions have been completed (approximately 48 hours after the final session)
Reporting Status: Not Posted

30. Other Pre Specified Outcome: Change in the Positive And Negative Syndrome Scale (PANSS) Score
Description: If participants have a co-morbid diagnosis of Schizophrenia, this clinician-rated assessment will be used to monitor symptoms.
Time Frame: After all stimulation sessions have been completed (approximately 48 hours after the final session)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: The day after treatment was completed, the participant was asked to complete a questionnaire regarding any adverse events during the week. (If any adverse events were evident to the researcher during the treatment week, a note was made and this was included in the final assessment to prevent under reporting of side-effects if the participant forgot about these events by the end of the 5 day treatment).
Groups:
- Dorsolateral Prefrontal Cortex (L-DLPFC): The accelerated theta burst stimulation protocol will be applied to the left dorsolateral prefrontal cortex (L-DLPFC)
  Accelerated theta burst stimulation: All participants will receive iTBS (intermittent theta burst stimulation) to the left DLPFC (if participants do not respond to L-DLPFC stimulation, they may be offered stimulation at the ACC). Stimulation intensity will be standardized at 80% of resting motor threshold (adjusted for cortical depth).
  Stimulation will be delivered using the Brainsway TMS system.
- Anterior Cingulate Cortex (ACC): The accelerated theta burst stimulation protocol will be applied to the anterior cingulate cortex (ACC)
  Accelerated theta burst stimulation: All participants will receive iTBS (intermittent theta burst stimulation) to the ACC. Stimulation intensity will be standardized at 80% of resting motor threshold (adjusted for cortical depth).
  Stimulation will be delivered using the Brainsway TMS system.
Arm/Group | Dorsolateral Prefrontal Cortex (L-DLPFC) | Anterior Cingulate Cortex (ACC)
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/2
Other Adverse Events (participants affected / at risk) | 7/20 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dorsolateral Prefrontal Cortex (L-DLPFC) (N=20) | Anterior Cingulate Cortex (ACC) (N=2)
Self-harm (Psychiatric disorders) | 1 | 0 — Determined not to be related to study participation.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dorsolateral Prefrontal Cortex (L-DLPFC) (N=20) | Anterior Cingulate Cortex (ACC) (N=2)
Headache (Nervous system disorders) | 2 | 1
Fatigue (General disorders) | 4 | 0
Anxiety (Nervous system disorders) | 0 | 1
Pain during stimulation (General disorders) | 1 | 1
Toothache (General disorders) | 1 | 0
Jaw pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Redness on forehead (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-12-13): https://cdn.clinicaltrials.gov/large-docs/17/NCT03601117/Prot_SAP_002.pdf
  • Informed Consent Form (2020-04-10): https://cdn.clinicaltrials.gov/large-docs/17/NCT03601117/ICF_003.pdf